CLINICAL TRIAL: NCT02701751
Title: Metabolic Adaptations to Chronic and Acute Exercise in Overweight Adults (ATX-Study)
Acronym: ATX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Professor, Movement Science; Director, Substrate Metabolism Laboratory, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00102522
Record Dates: First submitted 2016-01-21; First posted 2016-03-08 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise session (Other): Subjects will exercise at a moderate intensity for 60 minutes. There are no different arms in this study.
  Interventions: Other: Exercise session

INTERVENTIONS:
Other: Exercise session — A blood sample and fat biopsy will be obtained before and after the 60 minute moderate exercise session. There is no drug or device intervention in this study.

SUMMARY:
The primary purpose of this study is to examine the effects of chronic exercise training and an acute session of exercise on key risk factors associated with Metabolic Syndrome (e.g., glucose tolerance, blood lipid profile, and blood pressure) and alterations in subcutaneous adipose tissue structure and metabolic function in overweight adults.

DETAILED DESCRIPTION:
Subjects will be asked to complete the Substrate Metabolism Laboratory General Screening Questionnaire and American Heart Association Health/Fitness Questionnaire to determine if they are eligible to complete the preliminary testing procedures. If eligible, subjects will be asked to visit the Substrate Metabolism Laboratory to participate in the preliminary testing procedures (listed below) before participating in the experimental trial.

PRELIMINARY TESTING PROCEDURES:

* Blood pressure, height and weight measurements
* Body Composition Assessment (~20 min)
* Exercise Fitness Test (~10 min)
* Resting Metabolic Rate (RMR) measurement (~30 min)
* 3 hour Oral Glucose Tolerance Test (OGTT)

EXPERIMENTAL TRIAL:

The evening before the experimental trial, subjects will eat a standardized dinner meal and snack. The meal and snack must be eaten at specific times as indicated by the research staff. After eating the snack, subjects will need to fast (no food or beverages - besides water) overnight.

Participants who exercise regularly will be instructed to exercise exactly 3 days before the experimental trial, and then abstain from their exercise training program until after the study is complete.

In the morning, subjects will return to the Substrate Metabolism Laboratory. The research team will collect a blood sample from the subject's hand or forearm and a small sample of fat tissue in the subject's abdomen with a needle. Next, subjects will exercise on a treadmill at a moderate intensity for about 1 hour. Immediately after exercising the research team will collect a second blood sample. Subjects will remain in the laboratory for 1 hour after exercising, and then the research team will collect another blood and fat tissue sample. Upon completion of the experimental trial, subjects will be provided a snack before leaving the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 25-35 kg/m2
* Regular exercisers: (≥4 days/wk of aerobic exercise; 30-60min/session at moderate and vigorous intensities)
* Non-exercisers: no regularly planned exercise/physical activity
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Blood pressure > 140/90 mm Hg
* Pregnant or lactating
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
PPARg mRNA expression | change from baseline at 1 hour post exercise
  The study team will quantify the abundance of key adipogenic markers in adipose tissue biopsy samples
Cytokine abundance in adipose tissue | change from baseline at 1 hour post exercise
  The study team will measure cytokine proteins in adipose tissue

SECONDARY OUTCOMES:
Total Cholesterol | change from baseline at 1 hour post exercise
  Plasma concentrations of total- cholesterol will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States